CLINICAL TRIAL: NCT01843283
Title: Meaningful Activity Intervention for Persons With Mild Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1R21NR013755-01 (NIH)
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Family Caregivers; Intervention studies
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily Enhancement Meaningful Activity (DEMA) (Experimental): The group member will receive Self-management Toolkit and 6 bi-weekly individualized sessions, 2 face-to-face and 4 via telephone delivered by a trained intervener. DEMA will provide autonomy support by helping patients to identify and prioritize activities, classify needs and goals, generalize manageable solutions, engage in self-selected activities under family support, and self-evaluate failure and success or renew problem-solving as needed.
  Interventions: Behavioral: Daily Enhancement Meaningful Activity (DEMA)
- Information Support (IS) (Active Comparator): The IS group will receive 2 face-to-face meetings to receive an overview of what will happen in the study and an initial Alzheimer Association, educational brochure. Then they will receive 4 biweekly follow-up phone calls and have the opportunity to ask only questions related to the educational materials.
  Interventions: Behavioral: Information Support (IS)

INTERVENTIONS:
Behavioral: Daily Enhancement Meaningful Activity (DEMA)
  Arms: Daily Enhancement Meaningful Activity (DEMA)
Behavioral: Information Support (IS)
  Arms: Information Support (IS)

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility of and satisfaction with the revised DEMA and to estimate effect sizes for DEMA through incorporation of a comparison group. Specific aims are as follows:

Aim 1: Evaluate feasibility of the study for MCI patient/caregivers. Aim 2: Estimate effect sizes for DEMA on MCI patient and caregiver outcomes. Aim 3: Evaluate MCI patients and family caregivers' satisfaction with and perceptions of DEMA or IS.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) affects as many as 20% of older adults who are at a greater risk of developing Alzheimer's disease (AD). MCI involves functional decline that may include decrements in engagement in meaningful activities and one's own sense of confidence/mastery, and it is associated with depressive symptoms, poor satisfaction with family communication, and declining physical function. Existing interventions for MCI patients and caregivers often focus on a single problem, such as memory or physical activity and there are no available multi-faceted supportive care interventions to meet the needs of the MCI patients and their caregivers in order to prevent premature disengagement and risk for depressive symptoms. The Daily Enhancement of Meaningful Activity (DEMA) intervention uses a family dyadic, strengths-based, and positive health approach that builds on existing dyadic skills and values to accomplish meaningful activity engagement to address the priority needs for efficacious interventions to prevent premature disengagement and depressive symptoms in MCI patients. The DEMA builds on the investigators' previous descriptive work and gerontology theory, the model human occupation, and components of the Problem-Solving Therapy. The investigators' preliminary findings showed that the intervention and measures were acceptable, and suggestions were solicited from the participants for improving delivery. The purpose of this pilot study is to 1) evaluate the feasibility and satisfaction of the revised DEMA intervention; and 2) estimate effect sizes for the intervention through the incorporation of a comparison group. The MCI-caregiver dyads (n = 36 dyads) will be randomized to the DEMA or informational support groups; each group will receive 6 bi-weekly sessions (2 face-to-face and 4-phone delivered) with a trained intervener. The data from MCI patients and caregivers outcomes will be collected at pre-intervention, immediately (two weeks) post-intervention, and 3 months post-program evaluation. Descriptive statistics analysis will be used for satisfaction with and perception of the DEMA or informational support groups and general linear mixed models will be used to estimate the effect sizes of the intervention on the proximal and distal outcomes. Findings will inform the design of a subsequent R01 to: 1) test the efficacy of DEMA for MCI patient-caregiver dyads in a longitudinal randomized clinical trial; and 2) explore the costs/benefits of implementation. If it is found to be efficacious, DEMA has the potential to slow the rate of disability progression from MCI to AD and improve quality of life outcomes for patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

MCI patients:

1. are aged 60 years or older,
2. speak English,
3. have both caregiver-reported, clinically significant decline in cognition and clinician-detected or research based cognitive impairment on the standardized health exam
4. have at least one cognitive assessment score below the 7th percentile
5. have a normal range in performance of daily living tasks based on informant interview information indicating that impairment does not rise to the level of dementia.

Family caregivers:

1. are adults ≥ 21 years of age;
2. have primary responsibility for providing unpaid care to an MCI relative, along with monitoring safety and providing social support
3. are able to read and speak English
4. are oriented to persons, places, and time [having a 6-item Mini-Mental State Examination (MMSE) score of 4 or above]

Exclusion Criteria:

MCI patients and family caregivers will be excluded if:

1. the MCI patient or family caregiver has a diagnosed bipolar disorder or untreated schizophrenia;
2. the family caregiver has significant cognitive impairment that may hinder participation (6-item MMSE < 4)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Patient_Depression symptoms: Patient Health Questionnaire Depression Scale (PHQ-9) | Change in depression from baseline to immediately (two-week)- and 3 months post-intervention

SECONDARY OUTCOMES:
Patient_satisfaction with communication: The subscale of Communication and Affective Responsiveness | Change in satisfaction with communication from baseline to immediately (two-week)- and 3 months post-intervention
Patient_Physical Function: Alzheimer disease cooperative study activities of daily living inventory. | Change in physical function from baseline to immediately (two-week)- and 3 months post-intervention
Patient_Life satisfaction : Life Satisfaction Index for the Third Age-Short Form | Change in life satisfaction from baseline to immediately (two-week)- and 3 months post-intervention
Patient_Satisfaction with program: Satisfaction with Meaningful Activity Program Scale is adapted from the Caregiver Satisfaction Scale | It will be collected at 3 months post-program evaluation
Patient_ Meaningful activities engagement performance and satisfaction: Canadian Occupational Performance Measure & weekly log | Change in meaningful activities engagement performance and satisfactionfrom baseline to immediately (two-weeks)- and 3 months post-intervention
Patient_Sense of confidence: Confidence Scale | Change in sense of confidence from baseline to immediately (two-week)- and 3 months- post program
Caregiver_Depressive Symptoms: PHQ-9 | Change in depressive symptoms from baseline to immediately (two-week)- and 3 months post-program evaluation
Caregiver_ Caregiver life changes: Caregiving Outcomes Scale | Change in caregivign outcomes from baseline to immediately (two-week)- and 3 months post-post program
Caregiver_- Satisfaction with program: Satisfaction with Meaningful Activity Program Scale is adapted from the Caregiver Satisfaction Scale | It will be assessed at 3 months post-program evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Lu, PhD, Principal Investigator — IU School of Nursing
Locations (1):
- Indiana University School of Nursing, Indianapolis, Indiana, United States